CLINICAL TRIAL: NCT03822234
Title: A Prospective Multicenter Randomized Controlled Clinical Trial of Extraperitonealization for Prevention of Parastomal Hernia After Ileal Conduit
Brief Title: A Clinical Trial of Extraperitonealization for Prevention of Parastomal Hernia After Ileal Conduit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Director, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2018-104-01
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ileal conduit (Experimental): With our modified ileal conduit technique
  Interventions: Procedure: Modified ileal conduit
- Conventional ileal conduit (No Intervention): Conventional ileal conduit

INTERVENTIONS:
Procedure: Modified ileal conduit — Modified ileal conduit (Extraperitonealization)
  Arms: Modified ileal conduit

SUMMARY:
Many complications may occur after ileal conduit, with the incidence increasing with time after surgery. Nearly half of the complications are related to stoma and ureteroileal anastomosis. The investigators believe that the surgical technique is responsible for these complications, and therefore have devised a modified technique for creating the ileal conduit that should help prevent these complications after surgery. The investigators' retrospective study shows that modified surgical technique for ileal conduit urinary diversion appears to be effective for reducing early and late complications related to the stoma. Thus the investigators would like to perform a prospective multicenter randomized controlled clinical study to prove the investigators' results.

The investigators plan to enroll 104 patients, and randomizedly divide the participants into two groups, with one group 52 patients undergoing conventional ileal conduit, another group 52 patients undergoing modified ileal conduit.

DETAILED DESCRIPTION:
The ileal conduit (Bricker) has been used for urinary diversion for more than half a century. Widely accepted to be a simple and safe form of urinary diversion, it remains one of the most commonly used techniques for urinary diversion after radical cystectomy for bladder cancer. However, many complications may occur after ileal conduit, with the incidence increasing with time after surgery. Interestingly, nearly half of the complications are related to stoma and ureteroileal anastomosis. Among the complications, parastomal hernia is the most common. Female gender, low preoperative serum albumin level, high BMI or severe obesity, and prior laparotomy have been shown to be risk factors for parastomal hernia. But the mechanisms by which these variables lead to stoma related complications have not yet been fully elucidated. The investigators believe that the surgical technique is responsible for these complications, and therefore have devised a modified technique for creating the ileal conduit that should help prevent these complications after surgery. The investigators' retrospective study shows that modified surgical technique for ileal conduit urinary diversion appears to be effective for reducing early and late complications related to the stoma. Thus the investigators would like to perform a prospective multicenter randomized controlled clinical study to prove the investigators' results.

The investigators plan to enroll 104 patients, and randomizedly divide the participants into two groups, with one group 52 patients undergoing conventional ileal conduit, another group 52 patients undergoing modified ileal conduit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender not limited, life expectancy is greater than or equal to 24 months；
2. ECOG score of patients: 0-1；
3. Volunteer to participate in this study and sign the informed consent；
4. T2-T4a, N0-x,M0 invasive bladder cancer; High risk non-muscular invasive bladder cancer T1G3(high grade) tumor; Tis in which BCG therapy failed; Recurrent non-invasive bladder cancer; TUR and bladder perfusion were used for treatment of uncontrolled extensive papillary lesions and bladder non-urothelial carcinoma;
5. Major organ functions, such as liver, kidney, bone marrow, heart and other important organs, were not significantly abnormal: AST, ALT≤2.5 upper limit of normal value (ULN); Total bilirubin (TBIL)≤1.5 ULN; Albumin (ALB)≥25g/L; Serum creatinine (CRE)≤1.5 ULN; Leukocytes≥3.5*109/L, neutrophils≥1.5*109/L, hemoglobin≥90g/L, platelets≥80*109/L; Left ventricular ejection fraction (LVEF) ≥50%; Electrocardiogram showed no obvious abnormality or no clinical significance.

Exclusion Criteria:

1. A history of major middle and lower abdominal surgery;
2. Obese patients （BMI≥40kg/m2）;
3. Failure to receive regular follow-up review as required;
4. Severe cardiovascular disease;
5. History of immunodeficiency and organ transplantation；
6. History of severe central nervous system disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Incidence of parastomal hernia in 2 years | 2 years
  Incidence of parastomal hernia in 2 years

SECONDARY OUTCOMES:
Incidence of stomal retraction in 2 years | 2 years
  Incidence of stomal retraction in 2 years
Incidence of stomal stenosis in 2 years | 2 years
  Incidence of stomal stenosis in 2 years
Incidence of stomal prolapse in 2 years | 2 years
  Incidence of stomal prolapse in 2 years
Overall Survival | up to 2 years. From date of randomization until the date of first documented date of death from any cause, whichever came first, assessed up to 24 months
  Overall Survival
Disease-Free Survival | up to 2 years. From date of randomization until the date of first documented progression or recurrence or date of death from any cause, whichever came first, assessed up to 24 months
  Disease-Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No